CLINICAL TRIAL: NCT03251404
Title: Effects of Two Injury Prevention Exercise Programs on Performance and Neuromuscular Function in Youth Football
Brief Title: Effects of Injury Prevention Exercises on Performance and Neuromuscular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: The Swedish Research Council (Other Government); Region Östergötland (Other)
Responsible Party: Principal Investigator, Martin Hägglund, Associate professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHägglundPerformance
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Sport Injury; Adherence, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Two-armed cluster randomized parallel trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors (performance tests and neuromuscular function) blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Control original (Active Comparator): The Knee Control program exercise program will be performed during the warm-up to each football practice (at least twice per week) during the 12 week intervention period.
  Interventions: Other: Injury prevention exercise programs
- Knee Control+ (Experimental): The Knee Control+ is an extension of the original Knee Control exercise program offering a wider selection of exercises (to increase adherence) and more physically challenging exercises (adapted for athletes in the late teens and provide further stimuli to increase player performance and neuromuscular function). The program will be performed during the warm-up to each football practice (at least twice per week) during the 12 week intervention period.
  Interventions: Other: Injury prevention exercise programs

INTERVENTIONS:
Other: Injury prevention exercise programs — The two intervention programs contain exercises aiming to increase lower extremity strength, core stability, balance and neuromuscular function.

SUMMARY:
This study evaluates the effects of two different injury prevention exercise programs on sports-relevant performance tests and neuromuscular function in youth football players. Half of participants will receive education on an existing and previously tested exercise program, while the other half will receive education on a newly developed exercise program.

DETAILED DESCRIPTION:
Injury prevention exercise programs have been developed for a variety of sporting contexts and many have proven to be efficacious in preventing injuries. Adherence with the training may, however, be an issue and poor adherence may limit the preventive effect. If using the preventive exercise programs can be shown to improve sports-relevant performance this may motivate both coaches and players to use these programs, since the reduction in injury risk is harder to notice for the individual.

This study focuses on a Swedish injury prevention exercise program called Knee Control. The program has been found efficacious in preventing acute knee injuries in girls' adolescent football players in previous trials. We have found, however, that coaches often modify the Knee Control program to improve program fit and player buy-in among female youth football players. Careful changes must be made to the program since there is a risk of compromising the preventive effect and the effect on performance if the training dose is too low or if effective exercises are replaced with other exercises. We have therefore further developed the Knee Control program, to a Knee Control+ program, to support the coaches in the tailoring of the program to preserve the preventive effect and hopefully enhance performance effects. By introducing more variation with easier and more difficult exercises, pair-exercises, competitive and plyometric elements the new Knee Control+ program may better fit both the youngest and the oldest players, which in turn may facilitate fidelity with and maintenance of the program.

The aim of the study is to compare the neuromuscular and performance effects of the original Knee Control and the new Knee Control+ programs among youth female and male football players. A secondary aim is to study player and coach experiences of the programs and their fidelity with the training protocol.

Hypothesis: We expect similar effects of both programs, or superior effects of the Knee Control+ program, showing that the programs are compatible but the program adherence and fidelity being better with Knee Control+.

Methods: Eight youth football teams (4 boys, 4 girls, age 13-17 years) with approximately 120 players will be included in the study. Four teams will receive education about the Knee Control program and four teams about the Knee Control+ program. All coaches and two to three players per team will take part in a workshop at baseline where registered physiotherapists will give practical instructions of the intervention exercise programs. The workshops will also contain theoretical information about injuries in football and the background for either the Knee Control or the Knee Control+ programs. The attending coaches and players will be able to test all exercises and receive feedback about correct movement technique.

Outcomes: Football-relevant performance and neuromuscular function will be tested at baseline and after 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Football teams who have training at least twice per week
* Healthy players who can exert themselves maximally during testing

Exclusion Criteria:

* Teams who have used the Knee Control or a similar injury prevention exercise program on a regular basis the last year
* Players who cannot take full part in measurements due to illnesses or injuries

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Change in performance on the agility t-test (s) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in performance on the single-leg hop for distance (m) | Baseline and 12 weeks
Change in performance on drop vertical jumps as measured with knee separation distance (m) | Baseline and 12 weeks
Change in performance on the 505 agility test (s) | Baseline and 12 weeks
Change in performance on the side-hop test (n) | Baseline and 12 weeks
Change in performance on the 10 m sprint test (s) | Baseline and 12 weeks
Change in performance on the 20 m sprint test (s) | Baseline and 12 weeks
Change in performance on evaluation of lower extremity landing technique during the tuck jump test (points) | Baseline and 12 weeks
Coach baseline and follow-up experiences of injuries and of the Knee Control and Knee Control+ programs | Baseline and 12 weeks
Coach reported compliance and fidelity with the program protocol | At follow-up 12 weeks
Player baseline and follow-up experiences of injuries and of the Knee Control and Knee Control+ programs | Baseline and 12 weeks
Injuries that occur during the intervention period (number of injured players in each group) | At follow-up 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hägglund, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Division of physiotherapy, Department of Medical and Health Sciences, Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Study data (de-identified player performance test scores) may be available at request from the principal investigator

REFERENCES:
- [Derived] Lindblom H, Walden M, Hagglund M. Performance Effects with Injury Prevention Exercise Programmes in Male Youth Football Players: A Randomised Trial Comparing Two Interventions. Sports Med Open. 2020 Nov 23;6(1):56. doi: 10.1186/s40798-020-00282-7. PMID 33226542
- [Derived] Sonesson S, Lindblom H, Hagglund M. Performance on sprint, agility and jump tests have moderate to strong correlations in youth football players but performance tests are weakly correlated to neuromuscular control tests. Knee Surg Sports Traumatol Arthrosc. 2021 May;29(5):1659-1669. doi: 10.1007/s00167-020-06302-z. Epub 2020 Oct 8. PMID 33030610
- [Derived] Lindblom H, Walden M, Carlfjord S, Hagglund M. Limited positive effects on jump-landing technique in girls but not in boys after 8 weeks of injury prevention exercise training in youth football. Knee Surg Sports Traumatol Arthrosc. 2020 Feb;28(2):528-537. doi: 10.1007/s00167-019-05721-x. Epub 2019 Sep 20. PMID 31541293